CLINICAL TRIAL: NCT03420261
Title: Hemostasis Evolution During Fluid Loading in Abdominal Surgery. Effects of Fluid Choice: Saline Versus Hydroxyethyl Starch (HAEMO Study, an Ancillary Study of FLASH Trial)
Brief Title: Hemostasis Evolution During Fluid Loading in Abdominal Surgery. Effects of Fluid Choice: Saline Versus Hydroxyethyl Starch (HAEMO Study)
Acronym: HAEMO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-346; 2014-005578-84 (Other: 2014-005578-84)
Record Dates: First submitted 2017-09-05; First posted 2018-02-05 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Postoperative Morbidity; Postoperative Mortality; Hemostasis Change
Keywords: Goal-directed therapy; Fluid loading; Abdominal surgery; Postoperative morbidity; Postoperative mortality; Individualized goal-directed fluid therapy; Elective or emergency abdominal surgery; General Anesthesia; Moderate-to-high risk surgical patients
MeSH Terms: interventions — Saline Solution; Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crystalloid group (Active Comparator): individualized goal-directed fluid optimization (cardiac preload) by 250 ml boluses of 0.9% saline (up to a maximum of 30 ml/kg)
  Interventions: Biological: 0.9% saline
- Colloid group (Experimental): individualized goal-directed fluid optimization (cardiac preload) by 250 ml boluses of HES 130/0.4 (up to a maximum of 30 ml/kg, VOLUVEN ®, Fresenius Kabi)
  Interventions: Biological: HES 130/0.4

INTERVENTIONS:
Biological: 0.9% saline — Fluid administration
  Arms: Crystalloid group
Biological: HES 130/0.4 — Fluid administration
  Arms: Colloid group

SUMMARY:
The primary purpose of the study is to evaluate whether the type of fluid (0.9% saline or 6% Hydroxyethyl starch 130/0.4) in the context of an individualized goal-directed fluid therapy is associated with a difference in morbidity and mortality within the first 14 days in patients at moderate-to-high risk of postoperative complications after abdominal surgery.

Further investigation include the analysis of hemostasis modifications according to the fluid group during the first 7 days after abdominal surgery.

DETAILED DESCRIPTION:
Fluid administration is the mainstay treatment for suspected hypovolemia during surgery, but the effects of different crystalloid and colloid solutions on outcome remain poorly explored in surgical patients.

Two recent international multicenter studies (6S and CHEST studies) have shown that, compared to crystalloid solutions, the use of hydroxyethyl starch (HES) could be responsible for higher morbidity, especially renal failure, and mortality in ICU patients, thus leading to a recent restriction of their range of indications.

In contrast, in surgical patients, recent meta-analyses have concluded on the absence of difference in terms of mortality and postoperative renal failure between crystalloids and latest generation HES. Excessive fluid administration during surgery is associated with increased risk of postoperative morbidity, including renal dysfunction and mortality. It has been suggested that, compared with the volume-restoring effects of colloids, crystalloid use may require the administration of higher fluid volumes, which may contribute to poorer outcomes. In the surgical context, clinical trials and meta-analyses have shown that individualized goal-direct fluid administration can reduce postoperative morbidity. Although most GDT studies have used colloid solutions for fluid loading, the effects of the type of fluids are currently unknown and crystalloids are proposed for first-line therapy.

Moreover conflicting results on hemostatic effects of HES have been reported. HES have been associated with increased bleeding volume and transfusion requirements, especially in the ICU setting in septic patients. Perioperative use of HES was not associated with such findings. Biological effects of HES on hemostasis has barely been investigated and only by diluting plasma of healthy donors with HES.

The proposed Haemo multicenter study will be conducted to assess if the use of HES or crystalloid solutions during an individualized GDT contribute to biological hemostatic differences in patients at moderate-to-high risk of postoperative complications after abdominal surgery. As these fluids are widely used during surgery and because of current concerns about the risks related to the use of HES-based products in ICU patients, the trial will provide important data to clinicians involved in perioperative care and hemostasis.

ELIGIBILITY:
Inclusion Criteria:

* • - Undergo elective or emergency abdominal surgery under general anesthesia

  * With an estimated surgical duration greater than or equal to 2 hours
  * With moderate-to-high risk of postoperative complications defined by an AKI risk index≥ class 3, as defined by the presence of at least 4 of the following factors: age> 56 years, male gender, intraperitoneal surgery, active congestive heart failure, ascites, hypertension, emergency surgery, mild or moderate renal insufficiency, diabetes mellitus treated by oral or insulin therapy
  * Included in Clermont-Ferrand and Montpellier centers

Exclusion Criteria:

* • - Age <18 years

  * Preoperative acute heart failure
  * Preoperative acute coronary insufficiency
  * Preoperative severe renal failure (defined by creatinine clearance <30 ml/min or requiring renal replacement therapy)
  * Preoperative shock defined by the need for vasoactive amines
  * History of allergy with the use of 6% hydroxyethyl starch 130/0.4
  * Contraindication to the use of HES: sepsis, burnt patient, renal insufficiency or dialysis, cerebral hemorrhage, ICU patient , hypervolemia, lung edema, dehydration, severe hypernatremia or severe hyperchloremia, severe hepatic insufficiency, congestive heart failure, severe coagulopathy, organ transplant
  * Patient's or relative's refusal to participate
  * Parturient or breastfeeding woman
  * Protected major (guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07-22 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Prothombin Time | at day 1
  Evaluation of hemostasis parameters
Activated Cephalin TimeF | at day 1
  Evaluation of hemostasis parameters
Fibrinogen level and activity | at day 1
  Evaluation of hemostasis parameters
Von Willebrand factor | at day 1
  Evaluation of hemostasis parameters
Coagulation cascade | at day 1
  Evaluation of hemostasis parameters
Thrombin Generation test | at day 1
  Evaluation of hemostasis parameters
Fibrin Clot Permeability Test | at day 1
  Evaluation of hemostasis parameters

CONTACTS AND LOCATIONS:
Overall Officials: Thomas GODET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Puechal X, DeBandt M, Berthelot JM, Breban M, Dubost JJ, Fain O, Kahn JE, Lequen L, Longy-Boursier M, Perdriger A, Schaeverbeke T, Toussirot E, Sibilia J; Club Rhumatismes Et Inflammation. Tocilizumab in refractory adult Still's disease. Arthritis Care Res (Hoboken). 2011 Jan;63(1):155-9. doi: 10.1002/acr.20319. PMID 20740616
- [Background] Tournadre A, Dubost JJ, Soubrier M. Treatment of inflammatory muscle disease in adults. Joint Bone Spine. 2010 Oct;77(5):390-4. doi: 10.1016/j.jbspin.2010.04.007. Epub 2010 Jun 2. PMID 20627789
- [Background] Soubrier M, Mathieu S, Payet S, Dubost JJ, Ristori JM. Elderly-onset rheumatoid arthritis. Joint Bone Spine. 2010 Jul;77(4):290-6. doi: 10.1016/j.jbspin.2010.04.004. Epub 2010 May 31. PMID 20554241